CLINICAL TRIAL: NCT03806881
Title: Long Term Follow-up After Primary or Revision Shoulder Arthroplasty With a Patient- Specific Glenius Implant: A Prospective Cohort Study
Brief Title: Long Term Follow-up After Primary or Revision Shoulder Arthroplasty With a Patient- Specific Glenius Implant
Status: Enrolling by invitation | Type: Observational
Sponsor: Materialise (Industry)
Responsible Party: Sponsor
Other Study IDs: SMAT009
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Arthroplasty, Replacement, Shoulder; Glenoid Cavity; Osteoarthritis of the Shoulder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: Patients treated with a Glenius Glenoid Reconstruction System
  Interventions: Device: reversed glenoid prothesis

INTERVENTIONS:
Device: reversed glenoid prothesis — All patients will undergo a primary or revision arthroplasty with Glenius according to the routine practice at the investigation site and will be followed at specified visiting moments, during which radiological and clinical data will be gathered.
  Other Names: Glenius Glenoid Reconstruction system

SUMMARY:
This post-market follow-up study investigates improvement in clinical and radiological outcome after reversed total shoulder arthroplasty with the patient-specific Glenius Glenoid Reconstruction system

DETAILED DESCRIPTION:
The Glenius glenoid implant is a solution for patients who need a reversed glenoid reconstruction (primary or revision) because of a severely damaged glenoid associated with severe bone loss. In these cases, standard reconstruction of the glenoid is not possible because of the lack of body support of the glenoid rim or columns.

The Glenius implant is custom-made prothesis: during pre-operative planning, the implant is designed based on a detailed 3D CT analysis of the defect with special reference to bone quality and the anatomy of the bone deficient glenoid. Optimized screw fixation trajectories are defined for each individual patient, which accommodate screws that are positioned and angled towards the best bone stock available in the glenoid/coracoid/scapula with each specific patient. The surgeon provides feedback on the the design and orientation of the implant needed to achieve the optimal inclination of the head and the position & offset of the joint's centre of rotation.

Because Glenius is a relatively new product and only for use in specific and complex cases of severy glenoid erosion, follow-up data on the clinical and radiological outcome are scarce. With this study we aim to collect long-term clinical and radiological follow-up data for patients treated with Glenius in a uniform, standardized way.

ELIGIBILITY:
Inclusion Criteria:

* patients having primary or revision shoulder joint replacement with severe glenoid bone defects
* Patient is 18 years of age or older
* Patient can follow the Glenius system procedure that is standard of care
* Patient is willing to cooperate in the required post-operative therapy
* Patient has participated in the informed consent process and has signed the EC approved informed consent form

Exclusion Criteria:

* Pregnant patients
* Skeletally immature patients
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients having primary or revision shoulder joint replacement with severe glenoid bone defects caused by:(1) Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis, (2) Inflammatory degenerative joint disease such as rheumatoid arthritis or (3) Congenital malformations, posttraumatic deformities or removal of components during revision surgery
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in baseline Constant-Murley Score after surgery | 6 weeks, 3 months, 1 year, 2 year, 5 years after surgery
  The Constant-Murley score is a clinical outcome scale composed of a number of individual parameters, defining the level of pain, the ability to carry out the normal daily activities of the patient, mobility and strength of the arm. The scores range from 0 (worst clinical outcome) to 100 (best clinical outcome).

SECONDARY OUTCOMES:
Change in baseline Simple Shoulder Test (SST) after surgery | 6 weeks, 3 months, 1 year, 2 year, 5 years after surgery
  The SST is a function scale with 12 items, used to assess improvement in shoulder function after treatment interventions and to check the patient's ability to tolerate or perform 12 activities of daily living. The scores range from 0 (worst functional outcome) to 100 (best functional outcome).
Change in baseline Oxford Shoulder Score (OSS) after surgery | 6 weeks, 3 months, 1 year, 2 year, 5 years after surgery
  The OSS is a 12-item patient-reported outcome specifically designed and developed for assessing outcomes of shoulder surgery e.g. for assessing the impact on patients' quality of life of degenerative conditions such as arthritis and rotator cuff problems. The score ranges from 0 (no pain or functional impairement) to 60 (worst pain and functional impairement).
change in general health EQ5D score after surgery | 6 weeks, 3 months, 1 year, 2 year, 5 years after surgery
  EQ-5D is a standardized patient-reported outcome for measuring generic health status. The questionnaire has two components: a health state description measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. and a general evaluation of their overall health status using the visual analogue scale (EQ-VAS).
change in baseline pain score using Visual Analogue Scales (VAS) after surgery | 6 weeks, 3 months, 1 year, 2 year, 5 years after surgery
  The VAS pain score is a patient-reported evaluation of pain intensity on a Visual Analogue Scales (VAS) between 0 (no pain) and 100 (worst pain imaginable).
Translational deviation from planned implant position | 6 weeks after surgery
  translational deviation (in mm) of the implant position on post-operative shoulder CT scan when compared to the planned position on the pre-operative CT scan.
Rotational deviation from planned implant position | 6 weeks after surgery
  Rotational deviation (in degrees) of the implant position on post-operative shoulder CT scan when compared to the planned position on the pre-operative CT scan.
Translational deviation from initial implant position | 1 year after surgery
  translational deviation (in mm) on a shoulder CT scan 1 year after surgery, compared to the position on the post-operative CT scan.
Rotational deviation from initial implant position | 1 year after surgery
  Rotational deviation (in degrees) on a shoulder CT scan 1 year after surgery, compared to the position on the post-operative CT scan.
Scapular notching | 6 weeks, 3 months, 1 year, 2 years, 5 years after surgery
  scapular notching will be graded according to the Sirveaux classification system (2004) on a shoulder radiograph. The classification goes from 0 (no notching) to 4 (erosion over the inferior screw with extension under the baseplate)
Radiolucensies | 6 weeks, 3 months, 1 year, 2 years, 5 years after surgery
  Radiolucencies surrounding the glenoid component will be graded according to the system of Lazarus (Lazarus et al 2002) on a shoulder radiograph. The classification goes from 0 (no lucensies) to 5 (gross lucensies and radiographic loosening)
Heterotopic ossifications | 6 weeks, 3 months, 1 year, 2 years, 5 years after surgery
  periarticular heterotopic ossification (HO) will be scored according to a modified Brooker classification system of HO of the hip (Verhofste et al 2016) on a shoulder radiograph. The classification goes from 0 (no ossifications) to 3 (complete ankylosis of the shoulder)
rate of implant revision surgeries up to 5 years after surgery | up to 5 years after surgery
  Implant survival will be calculated by calculating the rate of implant revision surgeries up to 5 years after surgery.
Complication rate | up to 5 year after surgery
  the number and kind of (severe) adverse (device) events: device/shoulder related A(D)Es, SA(D)Es and device deficiencies that could have led to an SAE will be collected.

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (3):
  - AZ St-Elisabeth, Herentals
  - University Hospital Leuven - Traumatology, Leuven
  - University Hospital Leuven - Orthopedics, Leuven
- Sint-Maartenskliniek, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No